CLINICAL TRIAL: NCT07046078
Title: Pilot Study of FLAG-Ida Followed Immediately by Reduced-Intensity Allogeneic HCT for Adults Age 60 and Older With Newly Diagnosed Adverse-Risk AML or Other High-Grade Myeloid Neoplasm
Brief Title: Combination Chemotherapy (FLAG-Ida) Followed Immediately by Reduced-Intensity Total Body Radiation Therapy and Donor Hematopoietic Cell Transplant for the Treatment of Adults Age 60 and Older With Newly Diagnosed Adverse-Risk Acute Myeloid Leukemia or Other High-Grade Myeloid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125246; NCI-2025-02981 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020835 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-06-04; First posted 2025-07-01 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia of Ambiguous Lineage; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Stem Cell Transplantation; Specimen Handling; Biopsy; Cytarabine; fludarabine; Idarubicin; Peripheral Blood Stem Cell Transplantation; pegylated granulocyte colony-stimulating factor; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FLAG-Ida, TBI, HCT) (Experimental): Patients receive granulocyte colony-stimulating factor SC QD on days -9 to -4 or days -7 to -4 as clinically indicated, fludarabine IV over 30 minutes QD on days -8 to -4, cytarabine IV over 2 hours QD on days -8 to -4, and idarubicin IV over 60 minutes QD on days -8 to -6. Patients undergo TBI QD on days -1 and 0 or BID on day -1 or 0. Patients then undergo allogeneic HCT with unmodified peripheral blood stem cells IV on day 0 or 1 day after TBI as clinically indicated. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MUGA or ECHO during screening and as clinically indicated, undergo bone marrow biopsy and/or aspiration throughout the study and blood sample collection during follow up.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Idarubicin; Procedure: Multigated Acquisition Scan; Biological: Peripheral Blood Stem Cell; Other: Questionnaire Administration; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and/or aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and/or aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Peripheral Blood Stem Cell — Given IV
  Other Names: PBSC; Peripheral Blood Stem Cells; peripheral stem cell; Peripheral Stem Cells
Other: Questionnaire Administration — Ancillary studies
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given SC
  Other Names: Recombinant Colony-Stimulating Factor 3; rhG-CSF
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase II trial tests the safety, side effects, and how well combination chemotherapy with fludarabine, high-dose cytarabine, granulocyte colony-stimulating factor (G-CSF), and idarubicin (FLAG-Ida) followed immediately by reduced-intensity total body radiation therapy, called total body irradiation (TBI), and donor hematopoietic cell transplant (HCT) works in treating adults age 60 and older with newly diagnosed adverse-risk acute myeloid leukemia (AML) or other high-grade myeloid cancer. Despite advances in supportive care and the approval of more than 10 new drugs since 2017, the outcomes of older adults with adverse-risk acute myeloid leukemia and other high-grade myeloid cancers remains poor. Most patients are expected to die from their cancer or the consequences of treatment-related side effects. Donor HCT is a very important part of any curative-cancer treatment for these patients. However, while accepted as standard care for decades, this treatment exposes patients to long periods of drug-induced low blood cell counts and the problems associated with low blood counts, like infections and bleeding, which are associated with significant risk of chronic side effects and death. This study will use a different approach to the upfront curative-cancer treatment of older adults with an adverse-risk AML or other high-grade myeloid cancer. This study will use intense chemotherapy followed a few days later by lower-dose TBI and donor HCT. Chemotherapy drugs, such as idarubicin, fludarabine, high-dose cytarabine work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. G-CSF helps the bone marrow make more white blood cells in patients with low white blood cell count due to cancer treatment. This approach allows effective treatment of cancer cells and overall reduction of the period of low blood cells counts. This decreases the risk for problems associated with low blood counts, such as infection and chronic side effects. Decreasing these are important for older adults who undergo HCT. This treatment strategy may improve treatment outcomes by allowing more patients to successfully undergo donor HCT and reduce the risk of low blood cell counts and the problems associated with low blood counts. Giving chemotherapy followed immediately by reduced-intensity TBI and donor HCT may be safe, tolerable and/or effective in treating adults age 60 and older with newly diagnosed adverse-risk AML or other high-grade myeloid cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive granulocyte colony-stimulating factor subcutaneously (SC) once daily (QD) on days -9 to -4 or days -7 to -4 as clinically indicated, fludarabine intravenously (IV) over 30 minutes QD on days -8 to -4, cytarabine IV over 2 hours QD on days -8 to -4, and idarubicin IV over 60 minutes QD on days -8 to -6. Patients undergo TBI QD on days -1 and 0 or twice daily (BID) on day -1 or 0. Patients then undergo allogeneic HCT with unmodified peripheral blood stem cells IV on day 0 or 1 day after TBI as clinically indicated. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo multigated acquisition scan (MUGA) or echocardiography (ECHO) during screening and as clinically indicated, undergo bone marrow biopsy and/or aspiration throughout the study and blood sample collection during follow up.

After completion of study treatment, patients are followed up at days 28, 56 and 80, at months 3 and 6 and at years 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* PARTICIPANTS: Age ≥ 60 years. Adults age < 60 years are eligible if they are felt to be unsuitable candidates for myeloablative conditioning as per physician assessment
* PARTICIPANTS: Ability to understand and willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of potential study participants
* PARTICIPANTS: Newly diagnosed, untreated high-risk myeloid or mixed myeloid/lymphoid neoplasm:

  * Adverse-risk AML (using 2022 International Consensus Classification for disease categorization and 2022 European LeukemiaNet [ELN] criteria for molecular/cytogenetic risk assignment)
  * Acute leukemia of ambiguous lineage (using 2022 International Consensus Classification for disease categorization)
  * High-risk myelodysplastic neoplasm (MDS) (Molecular International Prognostic System [IPSS-M] moderate high, high, or very high, OR ≥ 10% blasts in blood or marrow)
  * High-risk chronic myelomonocytic leukemia (CMML) (clinical/molecular CMML-specific prognostic scoring system [CPSS-Mol] intermediate-2 or high, OR ≥ 10% blasts in blood or marrow)

    * Prior treatment of MDS or CMML with lower-intensity therapy (e.g., growth factors, erythropoiesis-stimulating agents, and lenalidomide) is permissible, but patients may not have received prior hypomethylating agents
* PARTICIPANTS: Disease not requiring immediate anti-neoplastic therapy (e.g., presenting with leukopenia or pancytopenia), defined as a clinical scenario in which delay of systemic leukemia-directed treatment would be unsafe. Supportive cytoreduction with hydroxyurea for transient disease control is allowed, and does not constitute immediate anti-neoplastic treatment
* PARTICIPANTS: Interest in pursuing allogeneic HCT
* PARTICIPANTS: Available caregiver
* PARTICIPANTS: Karnofsky score ≥ 70; Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* PARTICIPANTS: Bilirubin ≤ 2.5 x institutional upper limit of normal unless elevation is thought to be due to hepatic infiltration by myeloid neoplasm, Gilbert's syndrome, or hemolysis
* PARTICIPANTS: Serum creatinine ≤ 1.5 mg/dL
* PARTICIPANTS: Prior autologous HCT is permissible if > 6 months after planned HCT on this study
* PARTICIPANTS: Participants of child-bearing potential must be willing to employ two highly effective and acceptable forms of contraception 7 days before initiation of study treatment and for at least 12 months after HCT. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test during screening (within 2 weeks of treatment initiation, per Fred Hutch Cancer Center [FHCC] standard of care [SOC]), where WOCBP are defined as all female participants between 18-55 years of age, unless postmenopausal or with hysterectomy
* PARTICIPANTS: HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* PARTICIPANTS: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load
* PARTICIPANTS: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen, as determined by the investigator, are eligible for this trial
* DONORS: Patients must have an HLA-matched related donor, an HLA-matched or mismatched unrelated donor, or an HLA- haploidentical donor who meets standard Fred Hutchinson Cancer Center (FHCC) and/or National Marrow Donor Program (NMDP) or other donor center criteria for peripheral blood stem cell (PBSC) donation as follows:

  * HLA-matched related donor: related to the patient and genotypically or phenotypically identical for HLA-A, B, C, DRB1 and DQB1. Phenotypic identity must be confirmed by high-resolution typing
  * HLA-matched unrelated donor:

    * 10/10 matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
    * Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT. If the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive. A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
  * HLA-mismatched unrelated donor:

    * HLA-matching must be based on results of high resolution typing at HLA-A, -B, -C, -DRB1, and -DQ
    * Mismatched for a single allele without antigen mismatching at HLA-A, B, or C as defined by high resolution typing but otherwise matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
    * HLA class I HLA-A, -B, -C allele matched donors allowing for any one or two DRB1 and/or DQB1 antigen/allele mismatch
    * Donor/recipient HLA mismatching at loci for which the patient is homozygous is not allowed (isolated rejection vector)
  * HLA-haploidentical donor:

    * Donors must be haploidentical relatives of the patients. Donor-recipient compatibility will be tested through HLA typing at high resolution for the HLA loci (-A, -B, -C, -DRB1, -DQB1). Donor and recipient should share at least 5/10 HLA loci

      * Donor age ≥ 12 years
      * Donor weight ≥ 40 kg
      * Ability of donors younger than 18 years of age to undergo apheresis without use of a vascular access device. Vein check must be performed and verified by an apheresis nurse prior to arrival
      * Donor must meet the selection criteria as defined by the Foundation of the Accreditation of Cell Therapy (FACT) and will be screened per the American Association of Blood Banks (AABB) guidelines
    * In case of more than one available haploidentical donor, preference should be given to younger age
    * Since detection of anti-donor-specific antibodies (anti-DSA) is associated with higher graft rejection rate, patients will be screened for anti-DSA pre-transplant. Use of donors requiring desensitization treatment of the patient are not permissible

Exclusion Criteria:

* PARTICIPANTS: Active central nervous system (CNS) disease
* PARTICIPANTS: Decompensated congestive heart failure and/or uncontrolled arrhythmia and/or significant medical history of cardiac disease precluding allogeneic HCT
* PARTICIPANTS: Significant medical history of pulmonary disease and/or symptoms suggestive of pulmonary disease precluding allogeneic HCT
* PARTICIPANTS: Treatment with any other approved or investigational anti-leukemia agent(s) at the time of initiation of study treatment
* PARTICIPANTS: Concomitant illness associated with a likely survival of < 1 year
* PARTICIPANTS: Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with antimicrobials and/or controlled or stable. Patients with fever thought to be secondary to myeloid malignancy are eligible
* PARTICIPANTS: Known hypersensitivity or contraindication to receiving any of the study drugs used in this trial, including post-transplant cyclophosphamide (PTCy)
* PARTICIPANTS: Pregnancy or lactation
* PARTICIPANTS: Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants starting study treatment with FLAG-Ida within 42 days of the date of informed consent | Up to 42 days after informed consent
  Will evaluate the proportion of participants starting study treatment with FLAG-Ida within 42 days of the date of informed consent.

SECONDARY OUTCOMES:
Number of patients transplanted | Up to 2 years
  Will evaluate the number of patients transplanted.
Time from day of consent to day of allogeneic hematopoietic cell transplant (HCT) | From day of consent to day of allogeneic hematopoietic cell transplant (HCT)
  Will evaluate time from day of consent to day of allogeneic HCT.
Reasons for failure to undergo allogeneic transplantation (allo-HCT) | Up to 2 years following Screening enrollment
  Identified reasons for failure to undergo allogeneic transplantation (e.g., lack of suitable donor, complications of disease) will be systematically categorized and quantitatively reported.
Incidence of adverse events | From start of conditioning (Day -9) to study-defined neutrophil engraftment, or adversely, to graft failure
  Will evaluate the number of participants with non-hematologic adverse events ≥ grade 3. Will use the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for toxicity and adverse event reporting.
Neutrophil count recovery | Day 0 to study-defined neutrophil engraftment, or adversely, to graft failure.
  Will evaluate the time to neutrophil count recovery. The day of neutrophil recovery will be the 1st day of 2 consecutive days of absolute neutrophil count at or above 500/µL.
Platelet count recovery | Day 0 to study-defined platelet engraftment
  Will evaluate the time to platelet count recovery. Platelet engraftment will be defined as the first of 7 days of a platelet count > 20,000/µl without subsequent transfusions for 7 days.
Incidence of severe adverse events | From start of conditioning (Day -9) to study-defined neutrophil engraftment, or adversely, to graft failure
  Will evaluate the number of participants with any severe adverse event. Will use the NCI CTCAE version 5.0 for toxicity and adverse event reporting.
Non-relapse mortality (NRM) | Up to day 100 after HCT
  Will evaluate the number of participants experiencing NRM by day +100 after HCT.
Rate of CD3 chimerism | At day 80 (+/- 7 days)
  Will evaluate the rate of peripheral blood CD3 chimerism at day 80 (±7 days). Mixed or full donor chimerism will be evidence of donor engraftment.
  Full chimerism: > 95% donor CD3+ T cells. Mixed chimerism: the detection of peripheral blood donor T cells (CD3+) and granulocytes (CD33+) as a proportion of the total peripheral blood T cell and granulocyte population, respectively.
Rate of CD33 chimerism | At day 80 (+/- 7 days)
  Will evaluate the rate of peripheral blood CD33 chimerism at day 80 (±7 days). Mixed or full donor chimerism will be evidence of donor engraftment. Full chimerism: > 95% donor CD3+ T cells. Mixed chimerism: the detection of peripheral blood donor T cells (CD3+) and granulocytes (CD33+) as a proportion of the total peripheral blood T cell and granulocyte population, respectively.
Incidence of acute graft versus host disease (GVHD) | Up to day 100
  Will evaluate the cumulative incidence of grade 2-4 acute GVHD by day +100.
Incidence of chronic GVHD | Up to day 365
  Will evaluate the cumulative incidence of chronic GVHD requiring systemic immunosuppressive therapy by day +365.
Number of participants achieving complete remission or complete remission with incomplete hematologic recovery by day +42 | Up to day 42
  Will evaluate the number of participants achieving complete remission or complete remission with incomplete hematologic recovery by day +42. Will be determined by peripheral blood count and bone marrow evaluation and categorized according to the 2022 European LeukemiaNet criteria.
Measurable ("minimal") residual disease (MRD)-negativity | Up to day 42
  Will evaluate the number of participants achieving MRD-negativity by day +42. Will be determined by peripheral blood count and bone marrow evaluation and categorized according to the 2022 European LeukemiaNet criteria.
Relapse-free survival | At day 180
  Will evaluate relapse-free survival at day +180. Will be determined by peripheral blood count and bone marrow evaluation and categorized according to the 2022 European LeukemiaNet criteria.
Overall survival | At day 180
  Will evaluate overall survival at day +180.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Milano, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No